CLINICAL TRIAL: NCT01270126
Title: Treatment of Patients With Optic Neuropathy Using Transorbital Alternating Current Stimulation - a Randomized Trial
Brief Title: Trial of Alternating Current Stimulation in Optic Neuropathy
Acronym: SCT_optnerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: EBS Technologies GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Study leader, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBS_optnerve_SCT
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2013-12

CONDITIONS: Optic Nerve Diseases; Optic Nerve Injuries; Optic Neuropathies
Keywords: optic neuropathy; alternating current stimulation; vision recovery; restoration; plasticity
MeSH Terms: conditions — Optic Nerve Diseases; Optic Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rtACS (Verum condition) (Experimental): Repetitive transorbital alternating current stimulation (rtACS)
  Interventions: Device: Repetitive transorbital alternating current stimulation
- Sham stimulation (placebo condition) (No Intervention): A clicking sound was presented and the same electrode montage set-up was used during rtACS- and placebo-stimulation, except that placebo patients received no current (stimulator turned off)

INTERVENTIONS:
Device: Repetitive transorbital alternating current stimulation — Repetitive, transorbital alternating current stimulation (rtACS) was applied with a multi-channel device generating weak current pulses in predetermined firing bursts of 2 to 9 pulses. The amplitude of each current pulse was below 1000µA. Current intensity was individually adjusted according to how well patients perceived phosphenes, i.e. any sensation of flickering light in response to the rtACS stimulation.
  Other Names: EBS Alpha Synch
  Arms: rtACS (Verum condition)

SUMMARY:
Non-invasive brain stimulation can increase cortical excitability in the visual system, but it is not known if this is of clinical value. The investigators now assessed if repetitive, transcranial alternating current stimulation (rtACS) can improve visual field size in patients with optic nerve damage. The investigators hypothesized that rtACS would improve visual functions within the defective visual field sectors of the visual field (primary outcome measure).

DETAILED DESCRIPTION:
In a prospective, double-blind, randomized, placebo-controlled clinical trial 22 patients with optic nerve damage were randomly assigned to a rtACS- (n=12) or placebo-group (n=10). Visual field measures, visual acuity and EEG-recordings were collected before and after a daily 20-40min treatment for 10-days and at a 2-months-follow-up. Primary outcome measure was detection accuracy (DA) in defective visual field sectors of computer-based high resolution perimetry (HRP). Secondary outcome parameters included DA in static and kinetic perimetry, reaction time (RT) in HRP, visual acuity (VA), contrast vision, and EEG power spectra.

ELIGIBILITY:
Inclusion Criteria

* patients with optic nerve lesion
* stable visual field defect with residual vision
* lesion age at least 6 months

Exclusion Criteria

* heart pacemakers and any metal artefacts in head and truncus
* epileptic seizure within the last 3 years
* photosensitive epilepsy as determined by EEG
* mental diseases (schizophrenia etc.)
* unstable diabetes, diabetes causing diabetic retinopathy
* macular degeneration, maculopathy with decimal visual acuity below 0.4
* high blood pressure
* instable or high level of intraocular pressure (i.e. >27 mmHg)
* presence of an un-operated tumor anywhere in the body
* total blindness
* primary or secondary glaucoma
* pathological nystagmus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, PhD, Principal Investigator — University of Magdeburg
Locations (1):
- Institute of Medical Psychology, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sabel BA, Fedorov AB, Naue N, Borrmann A, Herrmann C, Gall C. Non-invasive alternating current stimulation improves vision in optic neuropathy. Restor Neurol Neurosci. 2011;29(6):493-505. doi: 10.3233/RNN-2011-0624. PMID 22124039
- See also: Study protocol as submitted (ethical proposal) - link "clinical trials" — http://www.med.uni-magdeburg.de/fme/institute/imp/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Assessed for eligibility (n=325)from local institutional database and upon response on announcements in local newspapers from Nov 2006 - Dec 2008.
  * Excluded (n=303): not meeting inclusion criteria (n=248), declined to participate (n=40), other reasons (n=15)
Groups:
- rtACS (Verum Condition): Repetitive transorbital alternating current stimulation (rtACS)
  Repetitive transorbital alternating current stimulation : Repetitive, transorbital alternating current stimulation (rtACS) was applied with a multi-channel device generating weak current pulses in predetermined firing bursts of 2 to 9 pulses. The amplitude of each current pulse was below 1000µA. Current intensity was individually adjusted according to how well patients perceived phosphenes, i.e. any sensation of flickering light in response to the rtACS stimulation.
Period: Overall Study
Arm/Group | rtACS (Verum Condition) | Sham Stimulation (Placebo Condition)
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rtACS (Verum Condition) | Sham Stimulation (Placebo Condition) | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (14.3) | 51.9 (17.3) | 52.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Germany | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Detection Accuracy (DA) Change in Percent Over Baseline Within Defective Visual Field Sectors
Description: Central visual fields were assessed with computer-based high-resolution perimetry (HRP). Based on such plots, areas of the visual field were characterized as intact, partially damaged or absolutely impaired (blind). Detection accuracy (DA) change in percent above baseline within defective visual field sectors was defined as the primary outcome criterion.
Time Frame: Outcome measures were assessed at initial diagnostics (baseline) and after 10 days stimulation at post diagnostics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | rtACS (Verum Condition) | Sham Stimulation (Placebo Condition)
Number analyzed (Participants) | 12 | 10
percent change | 24.75 (22.40) | 39.16 (25.26)

2. Secondary Outcome: Other Visual and EEG Parameters
Description: Secondary outcome parameters included DA in static and kinetic perimetry, reaction time (RT) in HRP, visual acuity (VA), contrast vision, and EEG power spectra.
Time Frame: Nov 2006 - Dec 2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were cutaneous sensations (tingling) under the stimulation electrodes and temporary sleeping difficulties
Arm/Group | rtACS (Verum Condition) | Sham Stimulation (Placebo Condition)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 7/12 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rtACS (Verum Condition) (N=12) | Sham Stimulation (Placebo Condition) (N=10)
cutaneous sensation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) — induced by electric current, felt as tingling
sleeping difficulties (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No